CLINICAL TRIAL: NCT03348176
Title: The What and How in Weaning: A Randomized Controlled Trial to Assess the Effects of Vegetable-exposure and Responsive Feeding on Vegetable Acceptance in Infants and Toddlers
Brief Title: Baby's First Bites: Promoting Vegetable Intake in Infants and Toddlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Leiden (Other)
Collaborators: Wageningen University (Other); Danone Global Research & Innovation Center (Industry); Nutricia, Inc. (Industry)
Responsible Party: Principal Investigator, Judi Mesman, Prof. dr. J. Mesman, Universiteit Leiden
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 057-14-002
Record Dates: First submitted 2017-11-09; First posted 2017-11-20 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Vegetable Acceptance in Early Childhood; Childhood Obesity; Childhood Overweight
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Investigators coding parental outcome measures of the study from videomaterial are masked for study-arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vegetable exposure (Experimental): Repeated exposure to a variety of vegetables from the start of complementary feeding
  Interventions: Other: Vegetable exposure
- VIPP-Feeding Infants (Experimental): Promotion of responsive feeding practices from the start of complementary feeding
  Interventions: Behavioral: VIPP-Feeding Infants
- Exposure + VIPP-FI (Experimental): Combination of repeated exposure to vegetables and promotion of responsive feeding practices
  Interventions: Other: Vegetable exposure; Behavioral: VIPP-Feeding Infants
- Control (Sham Comparator): Phone calls on development child with no information on complementary feeding
  Interventions: Other: Control

INTERVENTIONS:
Other: Vegetable exposure — Repeated exposure to variety of vegetables
  Arms: Exposure + VIPP-FI; Vegetable exposure
Behavioral: VIPP-Feeding Infants — Promoting responsive feeding practices
  Arms: Exposure + VIPP-FI; VIPP-Feeding Infants
Other: Control — Phone calls with mother about development of child, no advice on complementary feeding
  Arms: Control

SUMMARY:
Overweight and obesity in preschool children is more and more common and predicts overweight in later childhood and adulthood. A healthy eating pattern with many vegetables decreases the risk to develop overweight. As many food preferences are learned in the first years of life, teaching children to like vegetables from the very start of eating solid foods is essential. Starting baby's first bites of solid foods with vegetables instead of more sweet tastes like fruits may promote vegetable liking. Also, it is important that parents know how to feed their children: e.g., paying attention to whether the child is hungry or full is essential, as is not pressuring them to eat. What is yet unknown is which of these two are more important to promote, to facilitate vegetable liking in young children. Is starting with vegetables most important, or educating parents on their feeding-techniques? And is a combination of both most effective? This study tests which of three interventions is most effective to promote vegetable intake and liking in children up until the age of 3 years: a) a focus on the 'what' (starting with vegetables); b) a focus on the 'how' (listen to your child's cues while feeding); c) a focus on both the 'what' and the 'how'. These three groups will be compared to a control group receiving no advice on how to introduce solid foods on children's vegetable intake and liking.

DETAILED DESCRIPTION:
The weaning period in infancy is an important time for introducing healthy eating patterns that include vegetables to protect children against the development of overweight. There is evidence that it is important what weaning infants are offered: starting exclusively with vegetables is more successful for the promotion of vegetable acceptance than starting with fruits. There is also evidence that it is important how infants are weaned: responsive feeding characterised by sensitive responses to infant cues during feeding fosters healthy eating. However, the what and the how of infant weaning have never been experimentally tested in the same study to determine their relative importance for fostering vegetable acceptance, nor have they been combined to test whether a focus on both may be superior to each approach separately. This study employs a randomised controlled design testing the effectiveness of (a) a focus on the what in weaning, i.e., a vegetable-exposure intervention; (b) a focus on the how in weaning, i.e., an intervention to enhance responsive feeding; (c) a combined focus on what and how in weaning in an integrated intervention; (d) an attention-control group. Vegetable acceptance will be measured before and directly after the interventions when the child is 18 months of age, and when the child is 24 and 36 months of age. The proposed study is based on a unique integration of expert knowledge from the field of nutrition and the field of parenting, which will provide new insights into the mechanisms underlying the development of vegetable acceptance in infants, and ultimately the prevention of overweight.

ELIGIBILITY:
Inclusion Criteria:

First-time mothers of healthy term infants who report to have good reading and writing skills in the Dutch language

Exclusion Criteria:

* Medical problems in the infant that influence the ability to eat
* Major psychiatric problems in the mother, like depression
* Mothers who are not willing to start weaning exclusively with prepared vegetable/fruit purees from the Nutricia brand
* Mothers who are not willing for themselves and/or their infants to be video-taped

Ages: 4 Months to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 255 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in vegetable intake | Measured at child age of 4-6 months (prior to intervention), 18 months (directly after intervention) and at child age of 24 and 36 months (6 and 18 months follow-up)
  Intake of vegetables as measured by 3 days of 24hr recall electronic diaries (using the Compl-eat system developed at Wageningen University)
Change in vegetable liking | Measured at child age of 4-6 months (prior to intervention), 18 months (directly after intervention) and at child age of 24 and 36 months (6 and 18 months follow-up)
  Liking of vegetables as measured by questionnaire (Barends et al., 2013)
Child self-regulation of energy intake | Measured at child age of 18 months
  Measured experimentally; protocol designed for this study. In essence, children eat a meal at home until they are full, and after a short break are offered a variety of snacks. How much of the snacks they eat is a measure of child self-regulation of energy intake
Change in child self-regulation of energy intake | Measured at child age of 4-6 months (prior to intervention), 18 months (directly after intervention) and at child age of 24 and 36 months (6 and 18 months follow-up)
  Measured by the Child Eating Behavior Questionnaire

SECONDARY OUTCOMES:
Change in child eating behavior | Measured at child age of 4-6 months (prior to intervention), 18 months (directly after intervention) and at child age of 24 and 36 months (6 and 18 months follow-up)
  Measured with the Child Eating Behavior Questionnaire
Change in child anthropometrics | Measured at child age of 4-6 months (prior to intervention), 18 months (directly after intervention) and at child age of 24 and 36 months (6 and 18 months follow-up)
  Height and weight of child combined to report zBMI
Change in self-reported maternal feeding style | Measured at child age of 4-6 months (prior to intervention), 18 months (directly after intervention) and at child age of 24 and 36 months (6 and 18 months follow-up)
  Measured with Infant Feeding Style Questionnaire
Change in observed maternal feeding style | Measured at child age of 4-6 months (prior to intervention), 18 months (directly after intervention) and at child age of 24 and 36 months (6 and 18 months follow-up)
  Observed during family meals with an observation scale based on the Responsiveness to Child Feeding Cues Scale (Hodges et al.). Maternal responsiveness to child hunger cues (scale range 1 (very unresponsive) - 5 (very responsive); higher score is better) and pacing (scale range 1 ((almost) never adequate - 5 (almost) Always adequate; higher score is better) will be coded

CONTACTS AND LOCATIONS:
Overall Officials: Judi Mesman, PhD, Principal Investigator — Leiden University
Locations (2):
- Netherlands (2):
  - Leiden University, Faculty of Social Sciences, Education and Child Studies, Leiden
  - Wageningen University, Department of Agrotechnology and Food Sciences, Wageningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mueller C, Mars M, Zeinstra GG, Perenboom C, Forde CG, Jager G. Sowing the Seeds of Taste? A Novel Approach to Investigate the Impact of Early Sweet Exposure on Children's Dietary Taste Patterns from 12 to 36 Mo. J Nutr. 2025 May;155(5):1466-1473. doi: 10.1016/j.tjnut.2025.03.017. Epub 2025 Mar 18. PMID 40113172
- [Derived] van Vliet MS, Schultink JM, Jager G, de Vries JHM, Mesman J, de Graaf C, Vereijken CMJL, Weenen H, de Wild VWT, Martens VEG, Houniet H, van der Veek SMC. The Baby's First Bites RCT: Evaluating a Vegetable-Exposure and a Sensitive-Feeding Intervention in Terms of Child Health Outcomes and Maternal Feeding Behavior During Toddlerhood. J Nutr. 2022 Feb 8;152(2):386-398. doi: 10.1093/jn/nxab387. PMID 34791320
- [Derived] van der Veek SMC, de Graaf C, de Vries JHM, Jager G, Vereijken CMJL, Weenen H, van Winden N, van Vliet MS, Schultink JM, de Wild VWT, Janssen S, Mesman J. Baby's first bites: a randomized controlled trial to assess the effects of vegetable-exposure and sensitive feeding on vegetable acceptance, eating behavior and weight gain in infants and toddlers. BMC Pediatr. 2019 Aug 1;19(1):266. doi: 10.1186/s12887-019-1627-z. PMID 31370830
- See also: Trial website, including participant information and possibility to enroll — http://babyseerstehapjes.nl/